CLINICAL TRIAL: NCT05875961
Title: A Phase 1, Randomized, Observer-Blind, Multi-Center, Dose Ranging Study to Evaluate the Immunogenicity, Safety and Tolerability of Different Formulations of an Adjuvanted or Non-Adjuvanted Cell Culture-derived A/H2N3 Subunit Influenza Virus Vaccine in Healthy Subjects 18 Years and Above
Brief Title: Study to Evaluate Immunogenicity, Safety and Tolerability of Adjuvanted and Non-Adjuvanted H2N3 Influenza Vaccines in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V204_01
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Influenza, Human; Infections; Respiratory Tract Infections; Virus Diseases; Infection Viral
Keywords: Influenza; Vaccine; MF59; Adjuvant; H2N3
MeSH Terms: conditions — Influenza, Human; Infections; Respiratory Tract Infections; Virus Diseases | interventions — MF59 oil emulsion

STUDY DESIGN:
Intervention Model Description: Eligible subjects are randomized in an equal ratio to one of the 6 different treatment groups (formulations) and will receive two doses of the allocated H2N3c vaccine (adjuvanted or non-adjuvanted) at 3 weeks apart, ie, at Day 1 and Day 22.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of low dose A/H2N3c + standard dose MF59 adjuvant
  Interventions: Biological: Low dose A/H2N3c + standard dose MF59
- Group B (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of intermediate dose A/H2N3c + standard dose MF59 adjuvant
  Interventions: Biological: Intermediate dose A/H2N3c + standard dose MF59
- Group C (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of high dose A/H2N3c + standard dose MF59 adjuvant
  Interventions: Biological: High dose A/H2N3c + standard dose MF59
- Group D (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of high dose A/H2N3c non-adjuvanted
  Interventions: Biological: High dose A/H2N3c non-adjuvanted
- Group E (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of lowest dose A/H2N3c + high dose MF59 adjuvant
  Interventions: Biological: Lowest dose A/H2N3c + high dose MF59
- Group F (Experimental): Eligible subjects who have been randomized to receive two intramuscular vaccinations (3 weeks apart) of low dose A/H2N3c + high dose MF59 adjuvant
  Interventions: Biological: Low dose A/H2N3c + high dose MF59

INTERVENTIONS:
Biological: Low dose A/H2N3c + standard dose MF59 — Two intramuscular injections (3 weeks apart) of cell culture-derived MF59 adjuvanted H2N3 vaccine
  Arms: Group A
Biological: Intermediate dose A/H2N3c + standard dose MF59 — Two intramuscular injections (3 weeks apart) of cell culture-derived MF59 adjuvanted H2N3 vaccine
  Arms: Group B
Biological: High dose A/H2N3c + standard dose MF59 — Two intramuscular injections (3 weeks apart) of cell culture-derived MF59 adjuvanted H2N3 vaccine
  Arms: Group C
Biological: High dose A/H2N3c non-adjuvanted — Two intramuscular injections (3 weeks apart) of cell culture-derived non-adjuvanted H2N3 vaccine
  Arms: Group D
Biological: Lowest dose A/H2N3c + high dose MF59 — Two intramuscular injections (3 weeks apart) of cell culture-derived MF59 adjuvanted H2N3 vaccine
  Arms: Group E
Biological: Low dose A/H2N3c + high dose MF59 — Two intramuscular injections (3 weeks apart) of cell culture-derived MF59 adjuvanted H2N3 vaccine
  Arms: Group F

SUMMARY:
This Phase 1, randomized, observer-blind, dose-ranging clinical study is evaluating 6 different formulations of MF59-adjuvanted and non-adjuvanted H2N3 influenza vaccine. Approximately 600 healthy adult subjects are to be randomized into 1 of 6 possible treatment groups with 100 subjects per group, stratified by age group (born after or before 1968). Each subject will receive an influenza vaccine injection on Day 1 and Day 22. Subjects will be followed up for approximately 12 months after the second vaccine injection.

The primary immunogenicity analysis is based on the Day 1, Day 8, Day 22, Day 29, and Day 43 serology data. The primary safety analysis is based on solicited local and systemic adverse events (AEs) reported within 10 days after each vaccination, unsolicited AEs reported within 3 weeks after each vaccination, and serious AEs (SAEs), medically attended AEs (MAAEs), AEs leading to withdrawal from the study, and AEs of special interest (AESIs) reported throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18 years of age and older on the day of informed consent who were not born in 1968.
* Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures including follow-up.
* Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method, at least 30 days prior to informed consent, which they intend to use for at least 2 months after the last study vaccination.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to study entry and who do not plan to do so until 2 months after the last study vaccination.
* A body mass index (BMI) ≥35 kg/m2.
* Progressive, unstable, or uncontrolled clinical conditions as per investigator's assessment. Subjects must be stable and unchanged for a minimum of 3 months.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  1. Clinical conditions.
  2. Systemic administration of corticosteroids at a dose of ≥20 mg/day of prednisone or equivalent for more than 14 consecutive days within 90 days prior to informed consent. Topical, inhaled and intranasal corticosteroids are permitted. Intermittent use (one dose in 30 days) of intra-articular corticosteroids are also permitted.
  3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* History of any medical condition considered an adverse event of special interest (AESI).
* Received immunoglobulins with immunomodulating effects or any blood products within 180 days prior to informed consent.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Study personnel or immediate family or household member of study personnel.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
* Individuals who received any other vaccines (with the exception of COVID-19 vaccines) within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
* Receipt of any (investigational or licensed) COVID-19 vaccine within 14 days (non-replicating vaccines) or 28 days (replicating vaccines) prior to enrollment or plan to receive any COVID-19 vaccine within 14 days from study vaccination.
* A known history of Guillain-Barre Syndrome or other demyelinating diseases such as encephalomyelitis and transverse myelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of hemagglutination inhibition (HI) antibodies against homologous H2N3 strain - Day 1 | Day 1
  GMT (HI) prevaccination
GMT of HI antibodies against homologous H2N3 strain - Day 8 | Day 8
  GMT (HI) 1 week postvaccination 1
GMT of HI antibodies against homologous H2N3 strain Day 22 | Day 22
  GMT (HI) 3 weeks postvaccination 1
GMT of HI antibodies against homologous H2N3 strain - Day 29 | Day 29
  GMT (HI) 1 week postvaccination 2
GMT of HI antibodies against homologous H2N3 strain - Day 43 | Day 43
  GMT (HI) 3 weeks postvaccination 2
GMT of microneutralization (MN) antibodies against homologous H2N3 strain - Day 1 | Day 1
  GMT (MN) prevaccination
GMT of MN antibodies against homologous H2N3 strain - Day 8 | Day 8
  GMT (MN) 1 week postvaccination 1
GMT of MN antibodies against homologous H2N3 strain - Day 22 | Day 22
  GMT (MN) 3 weeks postvaccination 1
GMT of MN antibodies against homologous H2N3 strain - Day 29 | Day 29
  GMT (MN) 1 week postvaccination 2
GMT of MN antibodies against homologous H2N3 strain - Day 43 | Day 43
  GMT (MN) 3 weeks postvaccination 2
Geometric mean fold increase (GMFI) of HI antibodies against homologous H2N3 strain - Day 8 | Day 8
  GMFI (HI) 1 week postvaccination 1 compared to prevaccination
GMFI of HI antibodies against homologous H2N3 strain - Day 22 | Day 22
  GMFI (HI) 3 weeks postvaccination 1 compared to prevaccination
GMFI of HI antibodies against homologous H2N3 strain - Day 29 | Day 29
  GMFI (HI) 1 week postvaccination 2 compared to prevaccination
GMFI of HI antibodies against homologous H2N3 strain - Day 43 | Day 43
  GMFI (HI) 3 weeks postvaccination 2 compared to prevaccination
GMFI of MN antibodies against homologous H2N3 strain - Day 8 | Day 8
  GMFI (MN) 1 week postvaccination 1 compared to prevaccination
GMFI of MN antibodies against homologous H2N3 strain - Day 22 | Day 22
  GMFI (MN) 3 weeks postvaccination 1 compared to prevaccination
GMFI of MN antibodies against homologous H2N3 strain - Day 29 | Day 29
  GMFI (MN) 1 week postvaccination 2 compared to prevaccination
GMFI of MN antibodies against homologous H2N3 strain - Day 43 | Day 43
  GMFI (MN) 3 weeks postvaccination 2 compared to prevaccination
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Day 1 | Day 1
  % ≥1:40 (HI) prevaccination
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Day 8 | Day 8
  % ≥1:40 (HI) 1 week postvaccination 1
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Day 22 | Day 22
  % ≥1:40 (HI) 3 weeks postvaccination 1
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Day 29 | Day 29
  % ≥1:40 (HI) 1 week postvaccination 2
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Day 43 | Day 43
  % ≥1:40 (HI) 3 weeks postvaccination 2
Percentages of subjects with MN titers ≥1:40 against homologous H2N3 strain - Day 1 | Day 1
  % ≥1:40 (MN) prevaccination
Percentages of subjects with MN titers ≥1:40 against homologous H2N3 strain - Day 8 | Day 8
  % ≥1:40 (MN) 1 week postvaccination 1
Percentages of subjects with MN titers ≥1:40 against homologous H2N3 strain - Day 22 | Day 22
  % ≥1:40 (MN) 3 weeks postvaccination 1
Percentages of subjects with MN titers ≥1:40 against homologous H2N3 strain - Day 29 | Day 29
  % ≥1:40 (MN) 1 week postvaccination 2
Percentages of subjects with MN titers ≥1:40 against homologous H2N3 strain - Day 43 | Day 43
  % ≥1:40 (MN) 3 weeks postvaccination 2
Percentages of subjects with seroconversion by HI against homologous H2N3 strain - Day 8 | Day 8
  % seroconversion (HI) 1 week postvaccination 1, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Percentages of subjects with seroconversion by HI against homologous H2N3 strain - Day 22 | Day 22
  % seroconversion (HI) 3 weeks postvaccination 1, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Percentages of subjects with seroconversion by HI against homologous H2N3 strain - Day 29 | Day 29
  % seroconversion (HI) 1 week postvaccination 2, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Percentages of subjects with seroconversion by HI against homologous H2N3 strain - Day 43 | Day 43
  % seroconversion (HI) 3 weeks postvaccination 2, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Percentages of subjects with seroconversion by MN against homologous H2N3 strain - Day 8 | Day 8
  % seroconversion (MN) 1 week postvaccination 1, defined as a ≥4-fold increase in MN titer postvaccination in those with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with baseline titer <LLOQ
Percentages of subjects with seroconversion by MN against homologous H2N3 strain - Day 22 | Day 22
  % seroconversion (MN) 3 weeks postvaccination 1, defined as a ≥4-fold increase in MN titer postvaccination in those with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with baseline titer <LLOQ
Percentages of subjects with seroconversion by MN against homologous H2N3 strain - Day 29 | Day 29
  % seroconversion (MN) 1 week postvaccination 2, defined as a ≥4-fold increase in MN titer postvaccination in those with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with baseline titer <LLOQ
Percentages of subjects with seroconversion by MN against homologous H2N3 strain - Day 43 | Day 43
  % seroconversion (MN) 3 weeks postvaccination 2, defined as a ≥4-fold increase in MN titer postvaccination in those with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with baseline titer <LLOQ
Number and percentages of subjects reporting solicited local and systemic adverse events (AEs) - Day 1 through Day 10 | Day 1 through Day 10
  10 consecutive days postvaccination 1
Number and percentages of subjects reporting solicited local and systemic AEs - Day 22 through Day 31 | Day 22 through Day 31
  10 consecutive days postvaccination 2
Number and percentage of subjects reporting any unsolicited AEs | Day 1 through Day 43
  For 3 weeks following each vaccination
Number and percentage of subjects reporting serious AEs (SAEs), AEs leading to withdrawal, AEs of special interest (AESI) and medically attended AEs (MAAEs) | Day 1 through Day 387
  From vaccination until study completion

SECONDARY OUTCOMES:
GMT of ELLA titers as a measure of anti-neuraminidase (NA) immunogenicity | Day 1, Day 8, Day 22, Day 29, Day 43
  GMT (ELLA) prevaccination, 1 and 3 weeks postvaccination
GMFI of ELLA titers as a measure of anti-NA immunogenicity | Day 8, Day 22, Day 29, Day 43
  GMFI (ELLA) 1 and 3 weeks postvaccination compared to prevaccination
Percentage of subjects with ≥4-fold increase in ELLA titer as a measure of anti-NA immunogenicity | Day 8, Day 22, Day 29, Day 43
  % ≥4-fold increase (ELLA) 1 and 3 weeks postvaccination compared to prevaccination
GMT of HI antibodies against homologous H2N3 strain - Persistence | Day 202, Day 387
  GMT (HI) 6 and 12 months postvaccination 2
GMT of MN antibodies against homologous H2N3 strain - Persistence | Day 202, Day 387
  GMT (MN) 6 and 12 months postvaccination 2
GMT of ELLA titer as a measure of anti-NA immunogenicity- Persistence | Day 202, Day 387
  GMT (ELLA) 6 and 12 months postvaccination 2
GMFI of HI antibodies against homologous H2N3 strain - Persistence | Day 202, Day 387
  GMFI (HI) 6 and 12 months postvaccination 2 compared to prevaccination
GMFI of MN antibodies against homologous H2N3 strain - Persistence | Day 202, Day 387
  GMFI (MN) 6 and 12 months postvaccination 2 compared to prevaccination
GMFI of ELLA titer as a measure of anti-NA immunogenicity- Persistence | Day 202, Day 387
  GMFI (ELLA) 6 and 12 months postvaccination 2 compared to prevaccination
Percentages of subjects with HI titers ≥1:40 against homologous H2N3 strain - Persistence | Day 202, Day 387
  % ≥1:40 (HI) 6 and 12 months postvaccination 2
Percentages of subjects with MN titers ≥1:40, ≥1:80 and ≥1:160 against homologous H2N3 strain - Persistence | Day 202, Day 387
  % ≥1:40, ≥1:80 and ≥1:160 (MN) 6 and 12 months postvaccination 2
Percentages of subjects with seroconversion by HI against homologous H2N3 strain - Persistence | Day 202, Day 387
  % seroconversion (HI) 6 and 12 months postvaccination 2, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Percentages of subjects with seroconversion by MN against homologous H2N3 strain - Persistence | Day 202, Day 387
  % seroconversion (MN) 6 and 12 months postvaccination 2, defined as a ≥4-fold increase in MN titer postvaccination in those with prevaccination titer ≥LLOQ, or a postvaccination MN titer ≥4×LLOQ for subjects with baseline titer <LLOQ
Percentage of subjects with ≥4-fold increase in ELLA titer as a measure of anti-NA immunogenicity - Persistence | Day 202, Day 387
  % ≥4-fold increase (ELLA) 6 and 12 months postvaccination 2 compared to prevaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Science and Strategy, Study Chair — Seqirus
Locations (7):
- United States (3):
  - Meridian Clinical Research, Rockville, Maryland
  - Meridian Clinical Research, Lincoln, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
- Philippines (4):
  - West Visayas State University Medical Center, Iloilo City
  - Manila Doctors Hospital, Manila
  - Quirino Memorial Medical Center, Quezon City
  - Silang Specialists Medical Center, Silang

IPD SHARING:
Plan to Share IPD: Undecided